CLINICAL TRIAL: NCT05200845
Title: The Role of Altered Nutrient Partitioning in Food Reward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Alexandra DiFeliceantonio, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 21-964
Record Dates: First submitted 2021-12-17; First posted 2022-01-21 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Fat Meal Then High Carb Meal (Experimental): Participants will undergo exposure sessions with flavored beverage solutions containing sucrose first. Then, they will undergo exposure sessions with flavored beverages containing sucralose. Participants will undergo the high fat meal test session inside the metabolic chamber first. Then they will undergo the high carbohydrate test meal session.
  Interventions: Other: Conditioned Stimulus + (CS+): Flavored beverage solution with 75 calories of sucrose; Other: Conditioned Stimulus - (CS-): Flavored beverage solution with sweetness-matched sucralose; Other: High-Fat Test Meal Inside a Metabolic Chamber; Other: High-Carbohydrate Test Meal Inside a Metabolic Chamber; Other: fMRI Scan
- Conditioned Stimulus- (CS-) Then Conditioned Stimulus+ (CS+), and High Fat Meal Then High Carb Meal (Experimental): Participants will undergo exposure sessions with flavored beverage solutions containing sucralose first. Then, they will undergo exposure sessions with flavored beverages containing sucrose. Participants will undergo the high fat meal test session inside the metabolic chamber first. Then they will undergo the high carbohydrate test meal session.
  Interventions: Other: Conditioned Stimulus + (CS+): Flavored beverage solution with 75 calories of sucrose; Other: Conditioned Stimulus - (CS-): Flavored beverage solution with sweetness-matched sucralose; Other: High-Fat Test Meal Inside a Metabolic Chamber; Other: High-Carbohydrate Test Meal Inside a Metabolic Chamber; Other: fMRI Scan
- Conditioned Stimulus- (CS-)Then Conditioned Stimulus+ (CS+) and High Carb Meal Then High Fat Meal (Experimental): Participants will undergo exposure sessions with flavored beverage solutions containing sucralose first. Then, they will undergo exposure sessions with flavored beverages containing sucrose. Participants will undergo the high carbohydrate meal test session inside the metabolic chamber first. Then they will undergo the high fat test meal session.
  Interventions: Other: Conditioned Stimulus + (CS+): Flavored beverage solution with 75 calories of sucrose; Other: Conditioned Stimulus - (CS-): Flavored beverage solution with sweetness-matched sucralose; Other: High-Fat Test Meal Inside a Metabolic Chamber; Other: High-Carbohydrate Test Meal Inside a Metabolic Chamber; Other: fMRI Scan
- Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Carb Meal Then High Fat Meal (Experimental): Participants will undergo exposure sessions with flavored beverage solutions containing sucrose first. Then, they will undergo exposure sessions with flavored beverages containing sucralose. Participants will undergo the high carbohydrate meal test session inside the metabolic chamber first. Then they will undergo the high fat test meal session.
  Interventions: Other: Conditioned Stimulus + (CS+): Flavored beverage solution with 75 calories of sucrose; Other: Conditioned Stimulus - (CS-): Flavored beverage solution with sweetness-matched sucralose; Other: High-Fat Test Meal Inside a Metabolic Chamber; Other: High-Carbohydrate Test Meal Inside a Metabolic Chamber; Other: fMRI Scan

INTERVENTIONS:
Other: Conditioned Stimulus + (CS+): Flavored beverage solution with 75 calories of sucrose — Participants will consume flavored beverage solutions containing 75 calories of sucrose in 6 exposure sessions within 1 week. One exposure session will include pre- and post-consumption blood draws over a 2-hour period, and one exposure session will include indirect calorimetry measurement pre- and post-consumption. The other 4 exposure sessions will occur at specified times outside the laboratory sessions. Subjective ratings of internal state (i.e., hunger, fullness, and thirst) will be collected throughout each exposure. Subjective ratings of liking and wanting of each beverage will also be assessed.
Other: Conditioned Stimulus - (CS-): Flavored beverage solution with sweetness-matched sucralose — Participants will consume flavored beverage solutions sweetened with sucralose to match the sweetness of 75 calories of sucrose in 6 exposure sessions within 1 week. One exposure session will include pre- and post-consumption blood draws over a 2-hour period, and one exposure session will include indirect calorimetry measurement pre- and post-consumption. The other 4 exposure sessions will occur at specified times outside the laboratory sessions. Subjective ratings of internal state (i.e., hunger, fullness, and thirst) will be collected throughout each exposure. Subjective ratings of liking and wanting of each beverage will also be assessed.
Other: High-Fat Test Meal Inside a Metabolic Chamber — A high-fat test meal (60% fat, 20% carbohydrate) will be provided after a 1-hour baseline measurement of substrate oxidation during a 6-hour metabolic chamber stay. Postprandial substrate oxidation will be measured for 5 hours.
Other: High-Carbohydrate Test Meal Inside a Metabolic Chamber — A high-carbohydrate test meal (60% carbohydrate, 20% fat) will be provided after a 1-hour baseline measurement of substrate oxidation during a 6-hour metabolic chamber stay. Postprandial substrate oxidation will be measured for 5 hours.
Other: fMRI Scan — A subset of participants with BMI > 25 will be invited to complete an functional magnetic resonance imaging (fMRI) scan as a feasibility measure. fMRI scans will be performed while beverages (without calories) used during the intervention are delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids. Because this is feasibility-based measure, the outcome is a count of participants who completed this task.

SUMMARY:
Obesity remains a public health epidemic despite substantial advances in treatment strategies and therapies in the last decade. Effective strategies to support maintenance of improved metabolic health and reduced body weight are still needed.

Signals from the gut to the brain are important in regulating metabolism and energy balance and have been linked with food reward and preference in metabolically healthy individuals with normal body mass index. In particular, post-ingestive signaling related to glucose metabolism has been linked with food reward and preference. However, not much is known about how these gut and brain signals interact to influence eating behaviors in states of obesity or altered metabolic health. In addition, evidence in rodent models and human studies indicates obesity is associated with a blunted brain response to foods compared with normal body weight. However, whether altered nutrient utilization, termed metabolic inflexibility, influences the relationship between obesity and food reward has yet to be studied.

The overall objective of this proof-of-concept pilot study is to assess the feasibility of measuring reward response following a flavor-nutrient conditioning paradigm across the normal to obese body mass index (BMI) range and in states of altered metabolic health. The aims of this study are: 1) to determine whether differences in reinforcement learning/flavor-nutrient conditioning of carbohydrate can be measured across the body mass index range; and 2) to determine the feasibility of assessing metabolic flexibility and whether a relationship between metabolic flexibility and calorie-predictive reward can be detected.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 18.5-40 kg/m2
2. Not pregnant or planning to become pregnant during study participation
3. Residing in the Roanoke area and/or willing/able to attend sessions at the Fralin Biomedical Research Institute
4. Able to speak and write in English
5. Specific to fMRI scan only: BMI between 25-35 kg/m2

Exclusion Criteria:

1. Current inhaled nicotine use
2. History of alcohol dependence.
3. Current or past diagnosis of diabetes or thyroid problems.
4. Glycated hemoglobin (Hemoglobin A1C) >5.7%
5. Taking medications known to influence study measures (including antiglycemic agents, thyroid medications, sleep medications)
6. Active medical or neurologic disorder.
7. Recent change in body weight (gain or loss of > 5 lbs within the past 3 months)
8. Current shift work (typical pattern of work/activity overnight)
9. Previous weight loss surgery
10. Adherence to a special diet within the past 3 months (e.g., low-carb or ketogenic diet, exclusion of food groups/specific macronutrients, intermittent fasting, etc.)
11. Allergy to any food or ingredient included in the study diets, meals, or beverages
12. Currently pregnant or planning to become pregnant during study participation
13. Claustrophobia
14. Contraindications for MRI, including pacemaker, aneurysm clips, neurostimulators, cochlear or other implants, metal in eyes, regular work with steel, etc. (Note: This is an fMRI-specific exclusion criterion. Participants may be allowed to participate in all other study sessions and measures that do not involve fMRI.)
15. Contraindications for bioelectrical impedance analysis, specifically implanted devices

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at Virginia Tech Carilion, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 individuals were screened for eligibility between February 1, 2022 and May 1, 2023 in Roanoke, VA.
Pre-assignment Details: 16 of 20 participants were randomized. Of those not randomized, 3 did not meet inclusion criteria and 1 declined to participate.
Groups:
- Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Fat Meal Then High Carb Meal: Participants underwent exposure sessions with flavored beverage solutions containing sucrose first. Then, they underwent exposure sessions with flavored beverages containing sucralose. Participants underwent the high fat meal test session inside the metabolic chamber first. Then they underwent the high carbohydrate test meal session.
- Conditioned Stimulus- (CS-) Then Conditioned Stimulus+ (CS+), and High Fat Meal Then High Carb Meal: Participants underwent exposure sessions with flavored beverage solutions containing sucralose first. Then, they underwent exposure sessions with flavored beverages containing sucrose. Participants underwent the high fat meal test session inside the metabolic chamber first. Then they underwent the high carbohydrate test meal session.
- Conditioned Stimulus- (CS-) Then Conditioned Stimulus+ (CS+), and High Carb Meal Then High Fat Meal: Participants underwent exposure sessions with flavored beverage solutions containing sucralose first. Then, they underwent exposure sessions with flavored beverages containing sucrose. Participants underwent the high carbohydrate meal test session inside the metabolic chamber first. Then they underwent the high fat test meal session.
- Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Carb Meal Then High Fat Meal: Participants underwent exposure sessions with flavored beverage solutions containing sucrose first. Then, they underwent exposure sessions with flavored beverages containing sucralose. Participants underwent the high carbohydrate meal test session inside the metabolic chamber first. Then they underwent the high fat test meal session.
Period: Overall Study
Arm/Group | Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Fat Meal Then High Carb Meal | Conditioned Stimulus- (CS-) Then Conditioned Stimulus+ (CS+), and High Fat Meal Then High Carb Meal | Conditioned Stimulus- (CS-) Then Conditioned Stimulus+ (CS+), and High Carb Meal Then High Fat Meal | Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Carb Meal Then High Fat Meal
Started | 3 | 5 | 5 | 3
Completed | 2 | 3 | 2 | 3
Not Completed | 1 | 2 | 3 | 0
Not completed — stopped collecting pilot data for metabolic chamber | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Fat Meal Then High Carb Meal | Conditioned Stimulus- (CS-) Then Conditioned Stimulus+ (CS+), and High Fat Meal Then High Carb Meal | Conditioned Stimulus- (CS-) Then Conditioned Stimulus+ (CS+), and High Carb Meal Then High Fat Meal | Conditioned Stimulus+ (CS+) Then Conditioned Stimulus- (CS-), and High Carb Meal Then High Fat Meal | Total
Number analyzed (Participants) | 3 | 5 | 5 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (7.0) | 26.2 (5.8) | 30.0 (8.1) | 30.0 (6.7) | 29.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 1 | 9
  Male | 1 | 3 | 1 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 5 | 4 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 5 | 3 | 3 | 13
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 5 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Preference- Liking
Description: Subjective ratings of liking of flavors used in the intervention were assessed at baseline and after the intervention. The generalized Labeled Magnitude Scale will be used. The scale is anchored by descriptors of "Most Disliked Sensation Imaginable" and "Most Liked Sensation Imaginable" at the lower and upper ends, respectively. The score is determined by the place on the scale participants select (range of scale is 0-100). An increase in score from baseline to post-intervention indicates an increase in liking.
Time Frame: Baseline and at 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Conditioned Stimulus + (CS+); Conditioned Stimulus - (CS-): Participants complete behavioral preference tests for conditions at baseline and after the conditioning paradigm in a post-test. All participants complete all conditions in a cross-over design.
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 15 | 15
units on a scale | 6.5 (10.7) | 4.5 (13.0)

2. Secondary Outcome: Post-test Preference - Wanting
Description: Subjective ratings of wanting of flavors used in the intervention will be assessed at baseline and after the intervention. A Visual Analog Scale will be used. Participants select a place on the line that corresponds with their subjective rating, and the score is determined by the place selected (range of scores is 0-100). The line is anchored by polar opposite descriptors ("Do not want at all" and "Want very much"). An increase in score from baseline to post-intervention indicates and increase in wanting.
Time Frame: Baseline and at 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 15 | 15
units on a scale | 50.6 (120.) | 47.7 (10.2)

3. Secondary Outcome: Change in Preference- Wanting
Description: Ad libitum intake will be used as a measure of wanting in a post-test session. Participants will be provided each beverage used during the intervention and asked to drink as much or as little of them as they would like over a 30-minute period. Total beverage intake over 30 minutes is reported as the outcome.
Time Frame: 30-minute measurement
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 15 | 15
ml | 187.4 (152.2) | 147.3 (140.6)

4. Secondary Outcome: Change in Preference- Wanting
Description: Forced choice will be used as a measure of wanting in a post-test session. Participants will be provided each of the beverages used during the intervention and asked to choose 1 to take home with them. The outcome variable is a count of number of participants who chose each beverage condition during the forced choice test.
Time Frame: 5-minute measurement
Population: In the post-test session, participants are asked to choose between the CS+ and CS- beverage which they would like to take home in a forced choice test.
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 15 | 15
Participants | 9 | 6

5. Secondary Outcome: Blood Oxygen Level-dependent (BOLD) Response to Beverages
Description: In a post-test session, functional magnetic resonance imaging (fMRI) scans were performed while beverages (without calories) used during the intervention and a tasteless solution are delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids. Only participants with BMI > 25 were invited to complete this portion of the study, per our protocol. In total, participants receive the CS+, CS-, and tasteless (control) solutions 24 times over the course of 2 runs. Contrasts of interest are the blood oxygen level-dependent (BOLD) response of CS+>tasteless solution and CS->tasteless solution deliveries. Parameter estimates for these contrasts are extracted and reported. A positive outcome reflects greater whole-brain BOLD response for the CS condition compared with a tasteless solution.
Time Frame: 30-minute measurement that occurs during the post-test, approximately 4 weeks after the first study session
Population: The sample size is smaller for this measure due to the feasibility assessment nature of the measure. Only a subset of our recruited participants were invited to complete this measure. Only individuals with BMI > 25 were recruited for this portion of the study.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Conditioned Stimulus + (CS+): In a post-test, beverages (without calories) used during the intervention were delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids during functional magnetic resonance imaging (fMRI). Liquids delivered include the CS+ and CS- conditions (without calories) and a tasteless solution. Per our study protocol, the purpose of the fMRI scan is to assess feasibility, and only participants with BMI > 25 kg/m2 were asked to complete this portion of the protocol. Outcomes presented here are blood oxygen-level dependent (BOLD) response for contrasts of CS+>tasteless solution deliveries.
- Conditioned Stimulus - (CS-): In a post-test, beverages (without calories) used during the intervention were delivered through a custom manifold fitted to a head coil and connected to a pump system that allows precisely timed and measured delivery of liquids during functional magnetic resonance imaging (fMRI). Liquids delivered include the CS+ and CS- conditions (without calories) and a tasteless solution. Per our study protocol, the purpose of the fMRI scan is to assess feasibility, and only participants with BMI > 25 kg/m2 were asked to complete this portion of the protocol. Outcomes presented here are blood oxygen-level dependent (BOLD) response for contrasts of CS->tasteless solution deliveries.
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 6 | 6
arbitrary units | 0.0615 (0.1940) | 0.0467 (0.1025)

6. Secondary Outcome: Substrate Oxidation Response to Test Meals
Description: Indirect calorimetry in a metabolic chamber will be used to assess substrate oxidation response to high-fat and high-carbohydrate test meals.
Time Frame: 6-hour measurement
Population: Smaller sample size due to missing data
Measure: Mean (Standard Deviation); unit: fat oxidation grams/min*min
Groups:
- High Fat Test Meal: Participants underwent the high fat meal test session inside a metabolic chamber.
- High Carbohydrate Test Meal: Participants underwent the high carbohydrate meal test session inside a metabolic chamber.
Arm/Group | High Fat Test Meal | High Carbohydrate Test Meal
Number analyzed (Participants) | 12 | 7
fat oxidation grams/min*min | 4.6 (3.7) | -3.5 (3.3)

7. Secondary Outcome: Blood Glucose Response to Beverages
Description: Blood glucose will be assessed at baseline and at set time points for 1 hour after consumption of intervention beverages in one exposure session.
Time Frame: 2-hour measurement
Population: Smaller sample size due to missing data
Measure: Mean (Standard Deviation); unit: mg/dl*min
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 15 | 14
mg/dl*min | 882.4 (404.5) | 37.9 (315.6)

8. Secondary Outcome: Blood Insulin Response to Beverages
Description: Blood insulin will be assessed at baseline and at set time points for 2 hours after consumption of intervention beverages in an exposure session.
Time Frame: 2-hour measurement
Population: Smaller sample size due to missing data
Measure: Mean (Standard Deviation); unit: uIU/ml*min
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 15 | 14
uIU/ml*min | 694.4 (601.0) | 39.2 (132.9)

9. Secondary Outcome: Energy Expenditure in Response to Beverages
Description: Indirect calorimetry will be used to determine energy expenditure at baseline (for 30 minutes) and for 1 hour after consumption of intervention beverages in an exposure session.
Time Frame: 1.5-hour measurement
Population: Smaller sample size due to missing data
Measure: Mean (Standard Deviation); unit: kcal/min*min
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 14 | 12
kcal/min*min | 3.11 (2.97) | 0.76 (3.0)

10. Secondary Outcome: Respiratory Exchange Ratio in Response to Beverages
Description: Indirect calorimetry will be used to determine respiratory exchange ratio (RER) at baseline (for 30 minutes) and for 1 hour after consumption of intervention beverages in an exposure session. Areas under the curve for change in RER were calculated for each condition and presented as outcomes.
Time Frame: 1.5-hour measurement
Population: Smaller sample size due to missing data
Measure: Mean (Standard Deviation); unit: ratio*minutes
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 14 | 12
ratio*minutes | 2.9 (1.7) | 0.8 (1.3)

11. Secondary Outcome: Substrate Oxidation in Response to Beverages
Description: Indirect calorimetry will be used to determine substrate oxidation at baseline (for 30 minutes) and for 1 hour after consumption of intervention beverages in an exposure session.
Time Frame: 1.5-hour measurement
Population: Smaller sample size due to missing data
Measure: Mean (Standard Deviation); unit: carbohydrate oxidation grams/min*min
Arm/Group | Conditioned Stimulus + (CS+) | Conditioned Stimulus - (CS-)
Number analyzed (Participants) | 14 | 12
carbohydrate oxidation grams/min*min | 3.5 (2.0) | 0.9 (1.3)

ADVERSE EVENTS:
Time Frame: 7 weeks
Groups:
- Conditioned Stimulus+ (CS+): Participants underwent exposure sessions with flavored beverage solutions containing sucrose.
- Conditioned Stimulus- (CS-): Participants underwent exposure sessions with flavored beverage solutions containing sucralose.
Arm/Group | Conditioned Stimulus+ (CS+) | Conditioned Stimulus- (CS-) | High Fat Test Meal | High Carbohydrate Test Meal
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT05200845/Prot_SAP_000.pdf